CLINICAL TRIAL: NCT01716715
Title: A Randomized Phase II Study of NCI Supplied Cabozantinib (NSC #761968) Versus Weekly Paclitaxel (NSC #673089) in the Treatment of Persistent or Recurrent Epithelial Ovarian, Fallopian Tube or Primary Peritoneal Cancer
Brief Title: Cabozantinib or Paclitaxel in Treating Patients With Persistent or Recurrent Epithelial Ovarian, Fallopian Tube, or Primary Peritoneal Cavity Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02058; NCI-2012-02058 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); GOG-0186K; S13-00312; GOG-0186K (Other: NRG Oncology); GOG-0186K (Other: CTEP); U10CA180868 (NIH); U10CA027469 (NIH)
Record Dates: First submitted 2012-10-23; First posted 2012-10-30 (Estimated); Results first posted 2020-03-10 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-02

CONDITIONS: Recurrent Fallopian Tube Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Primary Peritoneal Carcinoma
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — cabozantinib; Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (cabozantinib-s-malate) (Experimental): Patients receive cabozantinib-s-malate PO QD on days 1-28.
  Interventions: Drug: Cabozantinib S-malate; Other: Laboratory Biomarker Analysis
- Arm II (paclitaxel) (Experimental): Patients receive paclitaxel IV over 1 hour on days 1, 8, and 15.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Paclitaxel

INTERVENTIONS:
Drug: Cabozantinib S-malate — Given PO
  Other Names: BMS-907351; Cabometyx; Cometriq; XL184
  Arms: Arm I (cabozantinib-s-malate)
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
  Arms: Arm II (paclitaxel)

SUMMARY:
This randomized phase II trial studies how well giving cabozantinib-s-malate or paclitaxel works in treating patients with persistent or recurrent epithelial ovarian, fallopian tube, or primary peritoneal cavity cancer. Cabozantinib-s-malate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. It is not yet known whether cabozantinib-s-malate or paclitaxel is more effective at treating patients with persistent or recurrent epithelial ovarian, fallopian tube, or primary peritoneal cavity cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the activity of cabozantinib (cabozantinib-s-malate) relative to weekly paclitaxel in patients with persistent or recurrent ovarian, fallopian tube, or primary peritoneal cancer with a log-rank test assessing progression-free survival (PFS) at 3.68 months (approximately pre-cycle 5) and 7.36 months (approximately pre-cycle 9).

SECONDARY OBJECTIVES:

I. To determine the frequency and severity of adverse events as assessed by Common Terminology Criteria for Adverse Events (CTCAE).

II. To estimate and compare the proportion of patients responding to therapy by Response Evaluation Criteria for Solid Tumors (RECIST), cancer antigen 125 (CA125) response, the overall survival (OS), and the duration of response in each arm.

TERTIARY OBJECTIVES:

I. To retrospectively correlate c-met proto-oncogene (MET) expression with overall outcome.

II. To retrospectively correlate c-MET copy number with overall outcome.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive cabozantinib-s-malate orally (PO) once daily (QD) on days 1-28.

ARM II: Patients receive paclitaxel intravenously (IV) over 1 hour on days 1, 8, and 15.

In both arms, courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have recurrent or persistent epithelial ovarian, fallopian tube or primary peritoneal carcinoma; histologic documentation of the original primary tumor is required via the pathology report
* Patients must have measurable disease or non-measurable (detectable) disease:

  * Measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded); each lesion must be greater than or equal to 10 mm when measured by computed tomography (CT), magnetic resonance imaging (MRI) or caliper measurement by clinical exam; or greater than or equal to 20 mm when measured by chest x-ray; lymph nodes must be greater than or equal to 15 mm in short axis when measured by CT or MRI
  * Non-measurable (detectable) disease is defined in this protocol as the absence of measurable disease but at least one of the following conditions:

    * Ascites and/or pleural effusion attributed to tumor
    * Solid and/or cystic abnormalities on radiographic imaging that do not meet RECIST 1.1 definitions for target lesions
* Patients with measurable disease must have at least one "target lesion" to be used to assess response on this protocol as defined by RECIST 1.1; tumors within a previously irradiated field will be designated as "non-target" lesions unless progression is documented or a biopsy is obtained to confirm persistence at least 90 days following completion of radiation therapy
* Patients must not be eligible for a higher priority Gynecologic Oncology Group (GOG) protocol, if one exists; in general, this would refer to any active GOG phase III or rare tumor protocol for the same patient population; in addition, patients must not be eligible for the currently active phase II cytotoxic protocol in platinum resistant disease
* Patients must have a GOG performance status of 0, 1, or 2
* Recovery from effects of recent surgery, radiotherapy, or chemotherapy to baseline or CTCAE =< grade 1 toxicity from all prior therapies except alopecia and other non-clinically significant adverse events (AE's):

  * Patients should be free of active infection requiring antibiotics (with the exception of uncomplicated urinary tract infection [UTI])
  * Any hormonal therapy directed at the malignant tumor must be discontinued at least one week prior to treatment
  * Any other prior therapy directed at the malignant tumor, including chemotherapy, biological/targeted (non-cytotoxic) agents and immunologic agents, must be discontinued at least three weeks prior to treatment
  * Chimeric or human or humanized monoclonal antibodies (including bevacizumab) or vascular endothelial growth factor (VEGF) receptor fusion proteins (including VEGF TRAP/aflibercept) must be discontinued for at least 12 weeks prior to treatment
  * Investigational agents must be discontinued for at least 28 days prior to treatment
  * Any prior radiation therapy must be discontinued at least four weeks prior to treatment
* Prior therapy

  * Patients must have had one prior platinum-based chemotherapeutic regimen for management of primary disease containing carboplatin, cisplatin, or another organoplatinum compound; this initial treatment may have included intraperitoneal therapy, consolidation, biologic/targeted (non-cytotoxic) agents (e.g., bevacizumab) or extended therapy administered after surgical or non-surgical assessment; if patients were treated with paclitaxel for their primary disease, this could have been given weekly or every 3 weeks
  * Patients are allowed to receive, but are not required to receive, two additional cytotoxic regimens for management of recurrent or persistent disease, with no more than 1 non-platinum, non-taxane regimen; treatment with weekly paclitaxel for recurrent or persistent disease is NOT allowed
  * Patients are allowed to receive, but are not required to receive, biologic/targeted (non-cytotoxic) therapy as part of their primary treatment regimen
  * Patients must have NOT received any biologic/targeted (non-cytotoxic) therapy targeting the VEGF and/or MET pathways for management of recurrent or persistent disease
  * For the purposes of this study, poly (adenosine diphosphate [ADP]-ribose) polymerase (PARP) inhibitors will be considered "cytotoxic"; patients are allowed to receive, but are not required to receive, PARP inhibitors for management of primary or recurrent/persistent disease (either alone or in combination with cytotoxic chemotherapy); PARP inhibitors will NOT count as a prior regimen when given alone
* Absolute neutrophil count (ANC) greater than or equal to 1,500/mcl
* Platelets greater than or equal to 100,000/mcl
* Hemoglobin greater than or equal to 9 g/dL
* Prothrombin time (PT) such that international normalized ratio (INR) is less than or equal to 1.3 x institutional upper limit of normal (ULN)
* Partial thromboplastin time (PTT) less than or equal to 1.3 x ULN
* Creatinine less than or equal to 1.5 x ULN
* Phosphorus, corrected calcium, magnesium and potassium greater than or equal to institutional lower limit of normal (LLN)
* Urine protein creatinine (UPC) ratio must be < 1.0 gm; if UPC ratio >= 1, collection of 24-hour urine measurement of urine protein is recommended
* Bilirubin less than or equal to 1.5 x ULN
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than or equal to 3 x ULN
* Alkaline phosphatase less than or equal to 2.5 x ULN
* Albumin greater than or equal to 2.8 g/dL
* Lipase less than or equal to 2 x ULN
* No radiologic or clinical evidence of pancreatitis
* Patients must have a normal baseline thyroid stimulating hormone (TSH); a history of hypothyroidism and/or hyperthyroidism is allowed
* Neuropathy (sensory and motor) less than or equal to grade 1
* Patients of childbearing potential must have a negative pregnancy test prior to the study entry and be practicing an effective form of contraception; sexually active subjects must agree to use medically accepted barrier methods of contraception (e.g., male or female condom) during the course of the study and for 4 months after the last dose of study drug, even if oral contraceptives are also used; all subjects of reproductive potential must agree to use both a barrier method and a second method of birth control during the course of the study and for 4 months after the last dose of study drug; pregnant women are excluded from this study
* Patients must have signed an approved informed consent and authorization permitting the release of personal health information
* Patients must meet pre-entry requirements

Exclusion Criteria:

* Patients who have had previous treatment with cabozantinib; patients who have received previous treatment with weekly paclitaxel for recurrent or persistent disease
* Patients with a history of other invasive malignancies, with the exception of non-melanoma skin cancer and other specific malignancies, are excluded if there is any evidence of other malignancy being present within the last three years; patients are also excluded if their previous cancer treatment contraindicates this protocol therapy
* Patients who have received prior radiotherapy to any portion of the abdominal cavity or pelvis or thoracic cavity within the last three years are excluded; prior radiation for localized cancer of the breast, head and neck, or skin is permitted, provided that it was completed more than three years prior to registration, and the patient remains free of recurrent or metastatic disease
* Patients who have received prior chemotherapy for any abdominal or pelvic tumor OTHER THAN for the treatment of ovarian, fallopian tube, or primary peritoneal cancer within the last three years are excluded; patients may have received prior adjuvant chemotherapy for localized breast cancer, provided that it was completed more than three years prior to registration, and the patient remains free of recurrent or metastatic disease
* Uncontrolled hypertension, defined as systolic greater than 140 mm Hg or diastolic greater than 90 mm Hg despite antihypertensive medications
* Myocardial infarction or unstable angina within 6 months prior to registration
* New York Heart Association (NYHA) class II or greater congestive heart failure
* History of serious ventricular arrhythmia (i.e., ventricular tachycardia or ventricular fibrillation) or serious cardiac arrhythmia requiring medication; this does not include asymptomatic atrial fibrillation with controlled ventricular rate
* Any history of congenital long QT syndrome
* The subject has a corrected QT interval calculated by the Fridericia formula (QTcF) > 500 ms within 28 days before randomization; note: if initial QTcF is found to be > 500 ms, two additional electrocardiogram (EKGs) separated by at least 3 minutes should be performed; if the average of these three consecutive results for QTcF is =< 500 ms, the subject meets eligibility in this regard
* Patients with serious non-healing wound, ulcer, or bone fracture within 28 days before treatment
* Patients with history of organ transplant
* Patients with active bleeding or pathologic conditions that carry high risk of bleeding, such as known bleeding disorder, coagulopathy, or tumor involving (in contact with, invading or encasing) major vessels
* Patients who have experienced any of the following:

  * Clinically-significant gastrointestinal bleeding within 6 months before the first dose of study treatment
  * Hemoptysis of >= 0.5 teaspoon (2.5 mL) of red blood within 3 months before the first dose of study treatment
  * Any other signs indicative of pulmonary hemorrhage within 3 months before the first dose of study treatment
* Patients who have radiographic evidence of cavitating pulmonary lesion(s)
* Patients who have tumor invading the gastrointestinal (GI) tract (esophagus, stomach, small or large bowel, rectum or anus), or any evidence of endotracheal or endobronchial tumor within 28 days before treatment
* Gastrointestinal disorders, particularly those with potential risk of perforation or fistula formation including:

  * Any of the following within 28 days of registration

    * Intra-abdominal tumor/metastases invading GI mucosa
    * Active peptic ulcer disease
    * Inflammatory bowel disease (including ulcerative colitis and Crohn's disease), diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis
    * Malabsorption syndrome
  * Any of the following within 6 months of registration

    * Abdominal fistula
    * Gastrointestinal perforation
    * Bowel obstruction or gastric outlet obstruction; note: patients requiring drainage gastrostomy (e.g., percutaneous endoscopic gastrostomy [PEG] tube) and/or parenteral hydration and/or nutrition are not eligible
    * Intra-abdominal abscess; note: complete resolution of an intra-abdominal abscess must be confirmed prior to registration even if the abscess occurred more than 6 months prior to registration
* Patients with history or evidence upon physical examination of central nervous system (CNS) disease, including primary brain tumor, seizures which are not controlled with non-enzyme inducing anticonvulsants, any brain metastases and/or epidural disease, or history of cerebrovascular accident (CVA, stroke), transient ischemic attack (TIA) or subarachnoid hemorrhage within six months prior to the first date of study treatment
* The subject requires chronic concomitant treatment of strong cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) inducers (e.g., dexamethasone, phenytoin, carbamazepine, rifampin, rifabutin, rifapentine, phenobarbital, and St. John's wort)
* Patients who are unable or unwilling to swallow tablets
* Patients who are pregnant or nursing
* The subject requires concomitant treatment, in therapeutic doses, with anti-coagulants such as warfarin or warfarin-related agents, heparin, thrombin or factor Xa inhibitors or antiplatelet agents (i.e. clopidogrel); low dose aspirin (=< 81 mg/day) low-dose warfarin (=< 1 mg/day) and prophylactic low molecular weight heparin are permitted
* Major surgery within 3 months of the first dose of cabozantinib if there were no wound healing complications or within 6 months of the first dose of cabozantinib if there were wound complications
* Minor surgery within 1 month of the first dose of cabozantinib if there were no wound healing complications or within 3 months of the first dose of cabozantinib if there were wound complications
* Patients with concurrent uncompensated hypothyroidism or thyroid dysfunction within 7 days before the first dose of study treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2012-11-06 (Actual); Primary Completion 2015-03-16 (Actual); Study Completion 2019-02-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ursula A Matulonis, Principal Investigator — NRG Oncology
Locations (173):
- United States (173):
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - John Muir Medical Center-Concord Campus, Concord, California
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Gynecologic Oncology Associates-Newport Beach, Newport Beach, California
  - University of Colorado Hospital, Aurora, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Sudarshan K Sharma MD Limited-Gynecologic Oncology, Hinsdale, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Saint Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic PC - Ames, Ames, Iowa
  - McFarland Clinic PC-Boone, Boone, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - McFarland Clinic PC-Jefferson, Jefferson, Iowa
  - McFarland Clinic PC-Marshalltown, Marshalltown, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Woman's Hospital, Baton Rouge, Louisiana
  - Maine Medical Center-Bramhall Campus, Portland, Maine
  - Maine Medical Center- Scarborough Campus, Scarborough, Maine
  - Union Hospital of Cecil County, Elkton, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - University of Massachusetts Memorial Health Care, Worcester, Massachusetts
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Saint Dominic-Jackson Memorial Hospital, Jackson, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Freeman Health System, Joplin, Missouri
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - NYU Winthrop Hospital, Mineola, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - New Hanover Regional Medical Center/Zimmer Cancer Center, Wilmington, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Clinic North-Fargo, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Summa Akron City Hospital/Cooper Cancer Center, Akron, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lancaster Radiation Oncology, Lancaster, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - The Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - Baylor All Saints Medical Center at Fort Worth, Fort Worth, Texas
  - Lyndon Baines Johnson General Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - PeaceHealth Medical Group PC, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Harrison Medical Center, Bremerton, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Skagit Valley Hospital Regional Cancer Care Center, Mount Vernon, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Northwest Hospital, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - Olympic Medical Cancer Care Center, Sequim, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Rockwood Cancer Treatment Center-DHEC-Downtown, Spokane, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Saint Joseph Medical Center, Tacoma, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington
  - HSHS Sacred Heart Hospital, Eau Claire, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Medical Center, Marshfield, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Ascension Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Ascension Saint Michael's Hospital, Stevens Point, Wisconsin
  - Saint Michael's Hospital, Stevens Point, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - Diagnostic and Treatment Center, Weston, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin

REFERENCES:
- [Derived] Gaitskell K, Rogozinska E, Platt S, Chen Y, Abd El Aziz M, Tattersall A, Morrison J. Angiogenesis inhibitors for the treatment of epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Apr 18;4(4):CD007930. doi: 10.1002/14651858.CD007930.pub3. PMID 37185961
- [Derived] Matulonis UA, Sill MW, Makker V, Mutch DG, Carlson JW, Darus CJ, Mannel RS, Bender DP, Crane EK, Aghajanian C. A randomized phase II study of cabozantinib versus weekly paclitaxel in the treatment of persistent or recurrent epithelial ovarian, fallopian tube or primary peritoneal cancer: An NRG Oncology/Gynecologic Oncology Group study. Gynecol Oncol. 2019 Mar;152(3):548-553. doi: 10.1016/j.ygyno.2018.12.008. Epub 2018 Dec 23. PMID 30587441

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 111 patients were enrolled from November 6, 2012 to May 5, 2014
Groups:
- Cabozantinib: Cabozantinib 60 mg oral daily continously
- Paclitaxel: Paclitaxel 80mg/m2 administered weekly on days 1, 8 and 15
Period: Overall Study
Arm/Group | Cabozantinib | Paclitaxel
Started | 57 | 54
Completed | 55 | 50
Not Completed | 2 | 4
Not completed — Never Treated | 2 | 4

BASELINE CHARACTERISTICS:
Population: Enrolled participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Cabozantinib | Paclitaxel | Total
Number analyzed (Participants) | 57 | 54 | 111
Age, Customized [Count of Participants; unit: Participants]
  20-29 years | 0 | 0 | 0
  30-39 years | 1 | 1 | 2
  40-49 years | 5 | 4 | 9
  50-59 years | 21 | 19 | 40
  60-69 years | 20 | 24 | 44
  70-79 years | 9 | 6 | 15
  >=80 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 54 | 111
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 4 | 2 | 6
  White | 50 | 48 | 98
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Event Free Survival
Description: Time from patient entry until progression, death, or beginning a subsequent therapy. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.",
Time Frame: The duration of time from study entry to time to progression or death,or begining a subsequent therapy, whichever occurs first, assessed up to 32 weeks
Population: Enrolled Patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cabozantinib | Paclitaxel
Number analyzed (Participants) | 57 | 54
months | 3.48 [2.79 to 4.07] | 4.96 [3.71 to 5.72]

2. Secondary Outcome: Number of Participants With Grade 3 or Higher Adverse Events by Type
Description: Toxicities will be characterized by their frequency and severity, grade 3 and above.
Time Frame: Up to 30 days after completion of study treatment
Population: Eligible and Treated participants
Measure: Count of Participants; unit: Participants
Groups:
- Grade 3 and Above on Cabozantinib: Grade 3 and above toxicities for participants on Cabozantinib 60 mg oral daily continously
- Grade 3 and Above on Paclitaxel: Grade 3 toxicities for participants on Paclitaxel 80mg/m2 administered weekly on days 1, 8 and 15
Arm/Group | Grade 3 and Above on Cabozantinib | Grade 3 and Above on Paclitaxel
Number analyzed (Participants) | 55 | 50
Participants
  Neutropenia | 2 | 4
  Anemia | 4 | 0
  Gastrointestinal | 15 | 2
  Metabolism/nutrition | 10 | 3
  Musculoskeletal/connective tissue | 1 | 0
  Nervous System | 3 | 0
  Renal/Urinary | 1 | 0
  Respiratory/thoracic/mediastinal | 3 | 1
  Skin/subcutaneous | 2 | 0
  Vascular disorders | 12 | 5

3. Secondary Outcome: Response, Assessed According to RECIST Version 1.1
Description: Complete and Partial Tumor Response by RECIST. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: CT or MRI used to follow lesion every 8 weeks for the first 8 months, then every 12 weeks until disease progression, approximately 2.5 years
Population: All enrolled participants
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Cabozantinib | Paclitaxel
Number analyzed (Participants) | 57 | 54
percentage of participants | 7.02 [2.4 to 15.3] | 24.07 [14.9 to 35.5]

4. Secondary Outcome: Percentage of Participants With CA125 Response.
Description: Complete and Partial Tumor Response by CA125. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.",
Time Frame: Prior to each cycle of treatment. Then follow-up every 3 months for 2 years then then every 6 months, up to 2.5 years.
Population: Participants evaluable by CA125
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Cabozantinib | Paclitaxel
Number analyzed (Participants) | 34 | 29
percentage of participants | 29.4 [16.9 to 44.8] | 58.6 [41.7 to 74.1]

5. Secondary Outcome: Overall Survival
Description: The time from randomization until death or date of last contact. Endpoint is death. Patients who are not observed with an endpoint are censored.
Time Frame: The duration of time from study entry to time of death or the date of last contact, an average of 2.5 years.
Population: All enrolled participants
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Cabozantinib | Paclitaxel
Number analyzed (Participants) | 57 | 54
months | 19.4 [12.3 to NA] — Upper limit of confidence interval has not been reached | NA [16 to NA] — The median and upper limit of confidence interval has not been reached

6. Secondary Outcome: To Estimate the Response Duration Among Patients Who Respond.
Description: The time participant is in response.Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.",
Time Frame: From the time measurement criteria are met for CR or PR until the first date that recurrent or progressive disease is objectively documented or date of death from any cause, whichever came first, assessed up to 18 months.
Population: Patients who respond.
Measure: Median (Full Range); unit: months
Arm/Group | Cabozantinib | Paclitaxel
Number analyzed (Participants) | 4 | 13
months | 3.8 [0.1 to 4.3] | 7.4 [3.5 to 16.7]

7. Other Pre Specified Outcome: c-Met Expression
Time Frame: Baseline
Reporting Status: Not Posted

8. Other Pre Specified Outcome: c-MET Copy Number
Time Frame: Baseline
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: During study treatment through 30 days after treatment ends, an average of 2.5 years.
Arm/Group | Cabozantinib | Paclitaxel
Serious Adverse Events (participants affected / at risk) | 25/55 | 8/50
Other Adverse Events (participants affected / at risk) | 55/55 | 50/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cabozantinib (N=55) | Paclitaxel (N=50)
Diarrhea (Gastrointestinal disorders) | 1 | 0
Small Intestinal Perforation (Gastrointestinal disorders) | 1 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 2 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 2
Mucositis Oral (Gastrointestinal disorders) | 1 | 0
Anal Pain (Gastrointestinal disorders) | 2 | 0
Ileal Obstruction (Gastrointestinal disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Fever (General disorders) | 0 | 2
Wound Complication (Injury, poisoning and procedural complications) | 2 | 0
Lipase Increased (Investigations) | 2 | 0
Aspartate Aminotransferase Increased (Investigations) | 1 | 0
Alanine Aminotransferase Increased (Investigations) | 2 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 2 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0
Neoplasms Benign, Malignant And Unspecified (Incl (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Memory Impairment (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Palmar-Plantar Erythrodysesthesia Syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Thromboembolic Event (Vascular disorders) | 4 | 2
Hypertension (Vascular disorders) | 2 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cabozantinib (N=55) | Paclitaxel (N=50)
Anemia (Blood and lymphatic system disorders) | 23 | 46
Sinus Bradycardia (Cardiac disorders) | 1 | 1
Palpitations (Cardiac disorders) | 2 | 0
Atrioventricular Block First Degree (Cardiac disorders) | 1 | 0
Cardiac Disorders - Other (Cardiac disorders) | 1 | 0
Ventricular Arrhythmia (Cardiac disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 4 | 3
Ear Pain (Ear and labyrinth disorders) | 3 | 1
Hypothyroidism (Endocrine disorders) | 12 | 0
Hyperthyroidism (Endocrine disorders) | 7 | 1
Endocrine Disorders - Other (Endocrine disorders) | 1 | 0
Watering Eyes (Eye disorders) | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 2
Blurred Vision (Eye disorders) | 3 | 5
Dry Eye (Eye disorders) | 0 | 1
Eyelid Function Disorder (Eye disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 7 | 1
Dry Mouth (Gastrointestinal disorders) | 10 | 0
Colitis (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 16 | 14
Enterovesical Fistula (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 37 | 19
Vomiting (Gastrointestinal disorders) | 20 | 5
Bloating (Gastrointestinal disorders) | 6 | 1
Abdominal Pain (Gastrointestinal disorders) | 21 | 13
Rectal Hemorrhage (Gastrointestinal disorders) | 4 | 4
Oral Dysesthesia (Gastrointestinal disorders) | 2 | 0
Obstruction Gastric (Gastrointestinal disorders) | 1 | 0
Mucositis Oral (Gastrointestinal disorders) | 21 | 6
Lower Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Disorders - Other (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Pain (Gastrointestinal disorders) | 1 | 1
Oral Pain (Gastrointestinal disorders) | 3 | 0
Abdominal Distension (Gastrointestinal disorders) | 4 | 3
Nausea (Gastrointestinal disorders) | 34 | 23
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 6 | 0
Rectal Pain (Gastrointestinal disorders) | 1 | 1
Esophagitis (Gastrointestinal disorders) | 1 | 0
Fecal Incontinence (Gastrointestinal disorders) | 1 | 0
Hemorrhoids (Gastrointestinal disorders) | 1 | 1
Ascites (Gastrointestinal disorders) | 6 | 3
Toothache (Gastrointestinal disorders) | 1 | 0
Esophageal Pain (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 3 | 1
Pain (General disorders) | 8 | 7
Localized Edema (General disorders) | 2 | 1
Irritability (General disorders) | 0 | 1
Injection Site Reaction (General disorders) | 0 | 1
Flu Like Symptoms (General disorders) | 0 | 1
Edema Trunk (General disorders) | 1 | 0
Non-Cardiac Chest Pain (General disorders) | 3 | 0
Edema Limbs (General disorders) | 6 | 9
Fatigue (General disorders) | 43 | 35
Fever (General disorders) | 3 | 5
Gait Disturbance (General disorders) | 0 | 1
Chills (General disorders) | 2 | 0
Allergic Reaction (Immune system disorders) | 0 | 1
Wound Infection (Infections and infestations) | 1 | 0
Upper Respiratory Infection (Infections and infestations) | 1 | 4
Tooth Infection (Infections and infestations) | 1 | 1
Stoma Site Infection (Infections and infestations) | 1 | 0
Skin Infection (Infections and infestations) | 1 | 0
Rhinitis Infective (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1
Otitis Media (Infections and infestations) | 0 | 1
Papulopustular Rash (Infections and infestations) | 1 | 1
Mucosal Infection (Infections and infestations) | 2 | 0
Esophageal Infection (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 3 | 1
Catheter Related Infection (Infections and infestations) | 0 | 1
Enterocolitis Infectious (Infections and infestations) | 0 | 1
Bladder Infection (Infections and infestations) | 1 | 0
Anorectal Infection (Infections and infestations) | 1 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1
Burn (Injury, poisoning and procedural complications) | 0 | 1
Bruising (Injury, poisoning and procedural complications) | 1 | 3
Weight Loss (Investigations) | 9 | 2
Weight Gain (Investigations) | 0 | 2
Serum Amylase Increased (Investigations) | 7 | 3
Platelet Count Decreased (Investigations) | 28 | 6
Lymphocyte Count Decreased (Investigations) | 1 | 4
Lipase Increased (Investigations) | 11 | 0
Inr Increased (Investigations) | 1 | 0
Ggt Increased (Investigations) | 1 | 0
Creatinine Increased (Investigations) | 7 | 5
Neutrophil Count Decreased (Investigations) | 25 | 28
Blood Bilirubin Increased (Investigations) | 7 | 0
White Blood Cell Decreased (Investigations) | 31 | 32
Aspartate Aminotransferase Increased (Investigations) | 34 | 6
Alkaline Phosphatase Increased (Investigations) | 21 | 8
Alanine Aminotransferase Increased (Investigations) | 30 | 4
Activated Partial Thromboplastin Time Prolonged (Investigations) | 2 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 16 | 3
Hyponatremia (Metabolism and nutrition disorders) | 9 | 5
Hypomagnesemia (Metabolism and nutrition disorders) | 27 | 19
Hypokalemia (Metabolism and nutrition disorders) | 15 | 5
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 15 | 6
Hypoalbuminemia (Metabolism and nutrition disorders) | 15 | 9
Hyperuricemia (Metabolism and nutrition disorders) | 1 | 0
Hypernatremia (Metabolism and nutrition disorders) | 1 | 2
Hypermagnesemia (Metabolism and nutrition disorders) | 2 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 5 | 12
Hypercalcemia (Metabolism and nutrition disorders) | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 4 | 2
Anorexia (Metabolism and nutrition disorders) | 25 | 7
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 4 | 7
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 10 | 7
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 6 | 0
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Chest Wall Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Buttock Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 9 | 6
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 5
Neoplasms Benign, Malignant And Unspecified (Incl (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tremor (Nervous system disorders) | 0 | 2
Peripheral Sensory Neuropathy (Nervous system disorders) | 13 | 28
Peripheral Motor Neuropathy (Nervous system disorders) | 2 | 3
Paresthesia (Nervous system disorders) | 1 | 1
Memory Impairment (Nervous system disorders) | 1 | 0
Movements Involuntary (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 14 | 8
Dysgeusia (Nervous system disorders) | 15 | 2
Dizziness (Nervous system disorders) | 11 | 2
Concentration Impairment (Nervous system disorders) | 0 | 1
Cognitive Disturbance (Nervous system disorders) | 1 | 0
Ataxia (Nervous system disorders) | 2 | 2
Akathisia (Nervous system disorders) | 0 | 1
Personality Change (Psychiatric disorders) | 0 | 1
Restlessness (Psychiatric disorders) | 0 | 2
Libido Decreased (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 8 | 11
Euphoria (Psychiatric disorders) | 2 | 0
Depression (Psychiatric disorders) | 9 | 6
Delirium (Psychiatric disorders) | 1 | 0
Confusion (Psychiatric disorders) | 2 | 0
Anxiety (Psychiatric disorders) | 7 | 5
Agitation (Psychiatric disorders) | 2 | 0
Urine Discoloration (Renal and urinary disorders) | 1 | 0
Urinary Urgency (Renal and urinary disorders) | 1 | 1
Urinary Tract Obstruction (Renal and urinary disorders) | 1 | 0
Urinary Retention (Renal and urinary disorders) | 1 | 0
Urinary Incontinence (Renal and urinary disorders) | 1 | 3
Urinary Tract Pain (Renal and urinary disorders) | 1 | 0
Urinary Frequency (Renal and urinary disorders) | 4 | 0
Renal Colic (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 2 | 1
Hemoglobinuria (Renal and urinary disorders) | 0 | 1
Hematuria (Renal and urinary disorders) | 3 | 0
Cystitis Noninfective (Renal and urinary disorders) | 0 | 1
Vaginal Hemorrhage (Reproductive system and breast disorders) | 2 | 2
Pelvic Pain (Reproductive system and breast disorders) | 3 | 2
Vaginal Discharge (Reproductive system and breast disorders) | 1 | 2
Respiratory, Thoracic And Mediastinal Disorders - (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Voice Alteration (Respiratory, thoracic and mediastinal disorders) | 7 | 0
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Sinus Disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Postnasal Drip (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 11 | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 13 | 7
Bronchial Obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Skin And Subcutaneous Tissue Disorders - Other (Skin and subcutaneous tissue disorders) | 1 | 0
Skin Ulceration (Skin and subcutaneous tissue disorders) | 0 | 1
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Rash Acneiform (Skin and subcutaneous tissue disorders) | 2 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 3
Palmar-Plantar Erythrodysesthesia Syndrome (Skin and subcutaneous tissue disorders) | 18 | 1
Pain Of Skin (Skin and subcutaneous tissue disorders) | 1 | 0
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 11 | 7
Skin Hypopigmentation (Skin and subcutaneous tissue disorders) | 4 | 0
Nail Loss (Skin and subcutaneous tissue disorders) | 0 | 3
Nail Discoloration (Skin and subcutaneous tissue disorders) | 0 | 5
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 1 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 5 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 11 | 31
Thromboembolic Event (Vascular disorders) | 6 | 3
Lymphedema (Vascular disorders) | 0 | 2
Hypotension (Vascular disorders) | 1 | 1
Hypertension (Vascular disorders) | 24 | 5
Hot Flashes (Vascular disorders) | 3 | 5
Hematoma (Vascular disorders) | 2 | 0
Flushing (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less